CLINICAL TRIAL: NCT00152789
Title: Oxygenation of the Prostate Gland: a Polarographic Electrode Study in Men Undergoing Prostate Biopsy.
Brief Title: Normal Prostate: Oxygenation of the Prostate Gland in Men Undergoing Prostate Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Dr. Michael Milosevic, Principal Investigator, University Health Network
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 01-0102-C
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2008-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: Oxygen measurement - Eppendorf machine

SUMMARY:
This study is based on previous observation that, in men with localized prostate cancer, non-cancerous prostate tissue is hypoxic, and on the known contribution of hypoxia to the progression of cancer. Patients undergoing diagnostic prostate biopsy with serum prostate specific antigen (PSA) less than 10ng/ml and who have given informed consent will have oxygen measurements of the prostate and peri-prostatic tissue taken with the Eppendorf electrode at the time of biopsy. The oxygenation of normal prostate tissue will be compared to that of cancerous prostate tissue. In men with negative biopsies, the prostate tissue oxygen measurements will be compared with the peri-prostatic tissue oxygen measurements.

ELIGIBILITY:
Inclusion Criteria:

* Men due to undergo sextant prostate biopsy
* Serum PSA <10 ng/ml

Exclusion Criteria:

* Previous diagnosis of prostate cancer
* Inability to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Median pO2 and HP5 will be analyzed according to the presence or absence of tumour on biopsy | 7 years

SECONDARY OUTCOMES:
Median pO2 and HP5 for the prostate gland in each patient with negative biopsy result will be compared with the median pO2 and HP5 for peri-prostatic tissue. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada